CLINICAL TRIAL: NCT00846885
Title: A Randomized, Two-Way, Single-Dose, Open-Label Study to Evaluate the Bioequivalence of a Test Tablet Formulation of Sumatriptan Succinate, (100mg), Compared to and Equivalent Dose of a Commercially Available Reference Drug Product (Imitrex®, GlaxoSmithKline, USA) in 28 Fed, Healthy, Adult Subjects.
Brief Title: Sumatriptan Succinate 100 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 04225
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sumatriptan Succinate
- 2 (Active Comparator)
  Interventions: Drug: Imitrex®

INTERVENTIONS:
Drug: Sumatriptan Succinate — 100 mg Tablet
  Arms: 1
Drug: Imitrex® — 100 mg Tablet
  Arms: 2

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of sumatriptan from a test formulation of Sumatriptan Succinate 100 mg Tablets versus the reference Imitrex® 100 mg Tablets under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Non-smoking (i.e. non-smoker or non-tobacco user for at least 90 days prior to pre-study medical screening) male or female within an age range of 18-40 years.
* Body Mass Index (BMI = weight/height2) greater than 19 kg/m2 and less than 26 kg/m2.
* Normal findings in the physical examination, vital signs (blood pressure between 100-140/60-90 mmHg, heart rate between 50-80 beats/min) and 12-lead ECG.
* Negative for drugs of abuse, nicotine, alcohol, hepatitis B-surface antigen, hepatitis C and HIV, and for female subjects, pregnancy (serum β-CG).
* No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides they are not clinically significant.
* Female subjects who are surgically sterile for at least six months or post-menopausal for at least one year, or who will avoid pregnancy prior to the study, during the study and up until one month after the end of the study.

Exclusion Criteria

* Known history of hypersensitivity to sumatriptan (e.g. Imitrex®, Imigran®) and/or related drugs such as almotriptan, naratriptan, rizatriptan and zolmitriptan
* Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, unless judged not clinically significant by the Principal Investigator or medical designate.
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness during the last four weeks prior to entry into this study.
* Presence of any significant physical or organ abnormality.
* Any subject with a history of drug abuse.
* Any history or evidence of psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator, or medical designate.
* Use of any prescription medication within 14 days preceding entry into this study.
* Use of any monoamine oxidase (MAO) inhibitor drugs such as phenelzine or tranylcypromine within 30 days preceding entry into this study.
* Use of over the counter (OTC) medication within seven days preceding entry into this study (except for spermicidal/barrier contraceptive products).
* Female subjects: use of oral contraceptives or contraceptive implants (such as Norplant®) within 30 days prior to drug administration or a depot injection of progestogen drug (e.g. Depo-Provera®) within one year prior to drug administration.
* Female subjects: presence of pregnancy or lactation.
* Any subject who has had blood drawn within 56 days preceding this study, taken during the conduct of any clinical study at a facility other than BCR, or within the lockout period specified by a previous study conducted at BCR.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* Any subject who has donated blood within 56 days preceding this study.
* Any subject who has participated as a plasma donor in a plasmapheresis program within seven days preceding this study.
* Significant or recent history of asthma (after 12 years of age).
* Any subject with a recent (less than one year) history of alcohol abuse.
* Known history of frequent headaches or migraines.
* Any subject with a parental or sibling history of heart attack or stroke that occurred under the age of 40 years.
* Intolerance to venipuncture.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08; Primary Completion 2004-09 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ziaee, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Sumatriptan) First: 100 mg Sumatriptan Tablets test product dosed in first period followed by 100 mg Imitrex® Tablets reference product dosed in the second period.
- Reference (Imitrex®) First: 100 mg Imitrex® Tablets reference product dosed in first period followed by 100 mg Sumatriptan Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Sumatriptan) First | Reference (Imitrex®) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Test (Sumatriptan) First | Reference (Imitrex®) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test (Sumatriptan) First | Reference (Imitrex®) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Sumatriptan) First | Reference (Imitrex®) First | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  Black | 3 | 7 | 10
  White | 11 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 12 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Sumatriptan): 100 mg Sumatriptan Tablets test product dosed in either period.
- Reference (Imitrex®): 100 mg Imitrex® Tablets reference product dosed in either period.
Arm/Group | Test (Sumatriptan) | Reference (Imitrex®)
Number analyzed (Participants) | 28 | 28
ng/mL | 80.334 (43.6) | 71.483 (32.193)
Statistical Analysis 1: Comparison: Test (Sumatriptan) vs Reference (Imitrex®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 110, 90% CI [103 to 117] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 12 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Sumatriptan) | Reference (Imitrex®)
Number analyzed (Participants) | 28 | 28
ng*h/mL | 305.374 (116.446) | 288.099 (109.217)
Statistical Analysis 1: Comparison: Test (Sumatriptan) vs Reference (Imitrex®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 106, 90% CI [102 to 111] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 12 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Sumatriptan) | Reference (Imitrex®)
Number analyzed (Participants) | 28 | 28
ng*h/mL | 314.996 (117.628) | 298.953 (111.361)
Statistical Analysis 1: Comparison: Test (Sumatriptan) vs Reference (Imitrex®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 105, 90% CI [101 to 110] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.